CLINICAL TRIAL: NCT06072508
Title: Prognostic Interest of Vasorin in Septic Shock
Acronym: VASO-SHOCK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Hospitalier Abbeville (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2023_843_0073
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Sepsis; Acute Kidney Injury
Keywords: vasorin; Sepsis; angiotensin II; Acute Kidney Injury
MeSH Terms: conditions — Sepsis; Acute Kidney Injury | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Blood sampling — Blood sampling (at day 0 and day 3) for Vasn, Angiotensin 2 and clotting markers.

SUMMARY:
In septic shock, the intensity and duration of low blood pressure can lead to a critical reduction in renal tissue perfusion and lead to the onset of more or less severe Acute Kidney Injury (AKI). Vasorin (Vasn) is a protein strongly expressed in large vessels and kidneys, whose functions are still poorly known. Previous experimental studies show that Vasn is associated with decreased Angiotensin II concentrations, a vessel contractility defect and early mortality.

The investigators hypothesize that Vasn (the potential direct regulator of blood pressure) would be an early biomarker predicting the severity of AKI post septic shock, which may be associated with mortality from septic shock or lead to longer-term Chronic Renal Failure (CKD).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Hospitalized in intensive care or medical resuscitation units.
* With a septic shock state defined by 2 mmol/l lactate sepsis, requiring vasopressors to maintain mean blood pressure 65 mmHg (despite adequate vascular filling).
* Whether or not they have developed AKI.
* Patient/family information and collection of non opposition

Exclusion Criteria:

* Patients with chronic respiratory failure.
* Pregnant women.
* Patients in palliative care.
* Information for the patient/someone close and collection of his opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
correlation between vasorin concentration at day 0 and mortality rate | day 0
correlation between vasorin concentration at day 3 and mortality rate | day 3

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No